CLINICAL TRIAL: NCT03927196
Title: The Program to Assess the Influence of Routing and Extended Statin Counseling of Patient With Cardiovascular Risk Factors on the Choice of Medicine and Treatment Compliance
Brief Title: Primary Prevention Program
Acronym: 3P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Center for Preventive Medicine (Other Government)
Collaborators: The League of Clinical Research, Russia (Other)
Responsible Party: Sponsor
Organization: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 03-01/18
Record Dates: First submitted 2019-02-12; First posted 2019-04-25 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Primary Prevention of Cardiovascular Disease
Keywords: primary prevention; cardiovascular risk; hyperlipidaemia; adherence
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- extended statin counseling group (Experimental): Extended statins counseling. Patients are handed out information leaflets on the correction of risk factors, SMS reminders.
  Interventions: Behavioral: extended counseling
- convetional statin counseling group (No Intervention): Сounseling on the prevention of cardiovascular diseases and the use of drugs for this purpose

INTERVENTIONS:
Behavioral: extended counseling — Patients are handed out information leaflets on the correction of risk factors, SMS reminders, extended statins counseling.
  Arms: extended statin counseling group

SUMMARY:
A systematic collection of retrospective and prospective data based on non-intervention patient observation, aimed to assess the risks, course and outcomes of a disease or a group of diseases:

* the retrospective part: database of patients with cardiovascular risks;
* the prospective part: observation of patients in the real medical practice

DETAILED DESCRIPTION:
The research program will have two parts:

Stage1: identification of patients with moderate, high and very high cardiovascular risks, not having diseases of atherosclerotic genesis and requiring lipid-lowering drugs.

Stage 2: a prospective observation of patients receiving primary medical prophylaxis of CVD with atorvastatin

ELIGIBILITY:
Inclusion Criteria:

Men and women 40-65 years old with the presence of:

* moderate cardiovascular risk (<5% but ≥1% on a SCORE scale) and cholesterol level LDL ≥3.0 mmol / l, in which the target is not reached during the improvement of lifestyle level of cholesterol-LDL, and the attending physician considers appropriate the appointment lipid-lowering drugs (statins), or
* high cardiovascular risk (≥5% but <10% on a SCORE scale) and cholesterol level LDL ≥ 2.5 mmol / l, or
* very high cardiovascular risk (≥10% on the SCORE scale) and cholesterol-LDL ≥1.8mmol / l, or
* atherosclerotic stenosis of the brachiocephalic arteries> 50% in the absence cerebrovascular diseases and the level of cholesterol-LDL ≥1.8 mmol / l, which do not have contraindications to taking statins and not taking drugs of this group in currently.

Exclusion Criteria:

* The presence of the following clinically significant events in anamnesis: myocardial infarction, stroke, myocardial infarction
* The presence of the following diseases at the time of statin administration: ischemic heart disease; heart failure; atherosclerotic disease of peripheral arteries; atherosclerotic stenosis of the brachiocephalic arteries in the presence of cerebrovascular disease; chronic renal failure with creatinine clearance <30 ml / min; liver disease with an increase in AST and ALT levels of more than 3 times, compared to the upper limit of normal; history of muscular or neuromuscular diseases, with elevated CPK; alcoholism, oncological, mental and other severe concomitant diseases; intolerance to statins in anamnesis; use of other lipid-modifying agents.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2912 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Change in the percentage of patients who achieved target LDL cholesterol level depending on the level of cardiovascular risk from baseline and 12 months | 12 months
  The primary objective of this study is to assess the influence of routing and extended statin counseling of patients with cardiovascular risk factors on the change in the percentage of patients who achieved target LDL cholesterol level from baseline through 12 months

SECONDARY OUTCOMES:
Assess the effect of routing and extended statin counseling on changes in treatment adherence | Baseline and Month 12
  The method used to measure adherence included the Morisky Medication Adherence Scale (MMAS - 4).
  Morisky Medication Adherence Scale is 4- item self-reported scale measuring medication taking behavior. Scores are transformed to a range of 0-4, in which higher scores reflect better adherence
Change from baseline in lipid levels (mmol/l) | Baseline, Month 3, Month 6 and Month 12
  To evaluate the impact of extended statin counseling on change of CVD risk factors (lipid levels) in patients with moderate, high and very high risk. Measurement of lipid levels at baseline and after 3,6,12 months
Change from baseline in blood pressure (mm Hg) | Baseline, Month 3, Month 6 and Month 12
  To evaluate the impact of standard and extended counseling on change of CVD risk factors (blood pressure). Measurement of blood pressure (mm Hg) at baseline and after 3,6,12 months
Impact of standard and extended counseling on statin therapy adherence | Baseline and Month 12
  The method used to measure adherence was KAP test. KAP test is the specially designed questionnaire for this study includes 14 questions, in patients with hyperlipidemia. KAP test summary score is an assessment of patients' knowledge about high cholesterol, their attitude to this problem and the application of this knowledge. Higher scores reflect better indicators of knowledge, attitudes and practices

CONTACTS AND LOCATIONS:
Overall Officials: Oxana M Drapkina, MD, PhD, Study Director — Director of National Medical Research Center for Preventive Medicine, Moscow
Locations (5):
- Russia (5):
  - Deputy Chief Medical Officer for Prevention at the Center for Medical Prevention, Astrakhan
  - Nizhny Novgorod Regional Center for Medical Prevention, Nizhny Novgorod
  - Regional Center for Medical Prevention, Novosibirsk
  - Samara Regional Center for Medical Prevention, Samara
  - Republican Center for Medical Prevention of the Republic of Bashkortostan, Ufa

IPD SHARING:
Plan to Share IPD: No